CLINICAL TRIAL: NCT05258396
Title: Exploring Cortical Remyelination in Children With Multiple Sclerosis
Acronym: REMYELIKIDS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APHP210916; 2021-A02792-39 (Other: IDRCB)
Record Dates: First submitted 2022-02-17; First posted 2022-02-28 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-03

CONDITIONS: Children With Multiple Sclerosis
Keywords: MRI; MS
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with MS (Experimental): Children with MS
  Interventions: Other: MRI without injection of contrast product
- Volunteers (Experimental): matched in age and sex with patients. Volunteers will perform only one brain MRI, as requested by the neurologist
  Interventions: Other: MRI without injection of contrast product

INTERVENTIONS:
Other: MRI without injection of contrast product — MRI without injection of contrast product

SUMMARY:
Multiple sclerosis (MS) in children, a rare disease, follows a relapsing remitting course with a shorter interval between the first 2 clinical events and higher annualized relapse rate as compared with MS in adults. Residual deficits following clinical events are less frequent. The vast majority of children and adolescents with MS are thought to have a greater potential for myelin repair than adults. However convincing data in the literature to support this hypothesis are lacking, because until now no imaging technique has been validated to measure remyelination in vivo.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) in children, a rare disease, follows a relapsing remitting course with a shorter interval between the first 2 clinical events and higher annualized relapse rate as compared with MS in adults. Residual deficits following clinical events are less frequent. The vast majority of children and adolescents with MS are thought to have a greater potential for myelin repair than adults. However convincing data in the literature to support this hypothesis are lacking, because until now no imaging technique has been validated to measure remyelination in vivo.

The investigator team has performed a first study to generate for the first time magnetization transfer ratio (MTR)-based maps of cortical myelin repair in 15 adult patients with MS. The team found that patients with MS showed a high variability in cortical myelin repair, with variable index of cortical remyelination. Moreover, there was a significant correlation between the index of cortical remyelination and clinical scores.

Even if childhood onset MS take longer to reach states of irreversible disability, severe disability will eventually occur at a young age. Moreover, pediatric MS could be responsible for cognitive disorders.

It is therefore of crucial relevance to develop research programs designed to generate novel imaging techniques to measure the efficacy of remyelinating therapies. Multiple sclerosis (MS) in children, a rare disease, follows a relapsing remitting course with a shorter interval between the first 2 clinical events and higher annualized relapse rate as compared with MS in adults. Residual deficits following clinical events are less frequent. The vast majority of children and adolescents with MS are thought to have a greater potential for myelin repair than adults. However convincing data in the literature to support this hypothesis are lacking, because until now no imaging technique has been validated to measure remyelination in vivo.

The team has performed a first study to generate for the first time magnetization transfer ratio (MTR) - based maps of cortical myelin repair in 15 adult patients with MS. The investigator team found that patients with MS showed a high variability in cortical myelin repair, with variable index of cortical remyelination. Moreover, there was a significant correlation between the index of cortical remyelination and clinical scores.

Even if childhood onset MS take longer to reach states of irreversible disability, severe disability will eventually occur at a young age. Moreover, pediatric MS could be responsible for cognitive disorders.

It is therefore of crucial relevance to develop research programs designed to generate novel imaging techniques to measure the efficacy of remyelinating therapies.

Finally, another extremely challenging issue in the care of children with MS is the difficulty of the transition between pediatric and adult care. Over last years, at the Pitié-Salpêtrière Hospital, the neurology team created a transition program called JUMP to improve medical, educational and psychosocial outcome for adolescent patients with MS .Taking part in the present study, young patients from 16 to 18 years old could have a direct access to the JUMP program, with the coordination of the dedicated nurses.

ELIGIBILITY:
Inclusion Criteria for patients :

* age between 12 years old and 18 years old
* RR-MS defined by 2017 McDonald criteria
* no relapse the last 4 weeks
* no methylprednisolone or prednisolone the last 4 weeks.
* affiliated to the social security system
* signature of the consent by the 2 holders of parental authority

Inclusion Criteria for Volunteers:

* age between 12 years old and 18 years old
* absence of any neurological
* signature of the consent by the 2 holders of parental authority

Exclusion Criteria for both groups:

* Parental rejection
* Contre-indication of brain MRI: pace maker, tatoo of the face, claustrophobia….
* Pregnancy, copper intrauterine device

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-08-11 (Actual); Primary Completion 2025-09-11 (Estimated); Study Completion 2025-09-11 (Estimated)

PRIMARY OUTCOMES:
MTR-based individual indices | 1 day
  To investigate the association between MTR-based individual indices of cortical myelin repair in children with MS and one cognitive score (Symbol Digital Modalities Test (SDMT)) at baseline

SECONDARY OUTCOMES:
indices of cortical remyelination | 6 months
  To investigate the association between individual indices of cortical remyelination and neurological disability

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Service de Neurologie Pédiatrique, Hôpital du Kremlin Bicêtre, Le Kremlin-Bicêtre
  - CIC Neurosciences - Pitié Salpêtrière, Paris
  - Service de Neurologie, GH Pitié Salpêtrière, Paris

IPD SHARING:
Plan to Share IPD: No